CLINICAL TRIAL: NCT02967341
Title: Validation of Central Venous (Port A Cath®) Blood Draws for Ciprofloxacin Pharmacokinetic Research in Patients Under Treatment for Childhood Cancer
Brief Title: Blood Draw Validation for Ciprofloxacin Pharmacokinetic Research in Pediatric Cancer Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Safepedrug-02
Record Dates: First submitted 2016-07-27; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-06

CONDITIONS: Childhood Cancer; Neutropenia
MeSH Terms: conditions — Neoplasms; Neutropenia | interventions — Ciprofloxacin; Vascular Access Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ciprofloxacin administration (Other): Blood will be drawn, in all participants, via Port A Cath and via a peripheral draw.
  Interventions: Other: Ciprofloxacin administration

INTERVENTIONS:
Other: Ciprofloxacin administration — Ciprofloxacin will be administered via the PAC directly followed by a NaCl 0.9% flush to wash the PAC. At least 1 hour afterwards 500 microliter of blood will be drawn via the PAC. Directly hereafter a blood draw of 500 microliter will be performed either via capillary blood sampling or via a venipuncture. If an anaesthesia is foreseen for another procedure (e.g. a lumbar puncture or an osseous punction), we will strive to perform the peripheral blood draw under anaesthesia.
  Other Names: Ciprofloxacin; Port A Cath (PAC)

SUMMARY:
To validate blood draws via a central venous catheter (Port A Cath ®) for pharmacokinetic studies of ciprofloxacin in patients under treatment for childhood cancer.

DETAILED DESCRIPTION:
The concentration of cipro will be determined using a validated high-performance liquid chromatographic (HPLC) method with fluorescence detection. Unbound concentration will be determined by adjusting the pH of the plasma samples to physiological pH (7.4) in a CO2 incubator, followed by ultrafiltration and extraction of ciprofloxacin from the ultrafiltrate (as described above) prior to injection onto the HPLC system.

ELIGIBILITY:
Inclusion Criteria:

Children who

* are between 1 month and 18 years of age
* are under treatment for any type of childhood cancer
* use ciprofloxacin for prophylaxis of febrile neutropenia as part of regular treatment
* have a PAC for intravenous medication and blood draws.

Exclusion Criteria:

Children will be excluded from this study if we are unable to

* obtain informed consent of both parents and assent of the child (if he/she is over 12 years of age)
* aspire blood from the PAC.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Correlation between ciprofloxacin concentration drawn via Port a Cath (PAC) versus capillary/venous punction | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Jutte van der Werff ten Bosch, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes